CLINICAL TRIAL: NCT06417450
Title: Utility of NESA Microcurrents in the Treatment of Sleep Disturbances, Disruptive Behaviours of Children With Autism Spectrum Disorders and in the Quality of Life of the Family Unit.
Brief Title: Usefulness of NESA Microcurrents in the Treatment of Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESATEA
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: physical therapy modality; sleep disorder; Quality of Life
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Intervention with electrical stimulation: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Intervention with electrical stimulation: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Placebo Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — Patients receive non-invasive neurostimulation through the Nesa device
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but electrical stimulation device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents.
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
The term or definition of Autism Spectrum Disorder (ASD) defines a pervasive neurodevelopmental disorder in which deficits in communication and social interaction, altered sensorimotor behaviours, repetitive, restricted and stereotyped interests and activities are observed.

One of the disorders most frequently associated with ASD, and which most affects the quality of life of the child and his or her family, is sleep disorders; it is estimated that between 50 and 80 percent of children with ASD present this alteration and generally continue to suffer from it in adolescence and adulthood; It has also been observed that there is a correlation between sleep problems and an increase in aggressive behaviour, social and emotional deficits and deficits in activities of daily living, which severely affects the child and his or her close family environment; they become emotionally destabilised in a notorious way, and this has a negative impact on their work and productive environment.

The microcurrents generated by the non-invasive neuromodulation device introduce, by means of a non-invasive technique (surface electrodes), electrical energy to normalise the nervous stimulus. This makes it an excellent complementary treatment to the activity of rehabilitation treatment. Its effects are achieved by establishing several input nerve pathways corresponding to the body's dermis, through which the signals are intellectualised in time-space. These signals are the basis for achieving normalisation of the nerve impulse by means of microcurrents.

DETAILED DESCRIPTION:
The main objective will be to test the influence of surface neuromodulation applied NESA on sleep disturbances in children with Autism Spectrum Disorders and how this is related to disruptive behaviours and quality of life in the family environment.

It is estimated to take 8 months from the design, management and development of the project, and does not have sources of funding.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of Autistic Spectrum Disorder, attending school in the City of San Juan de Dios in Las Palmas de Gran Canaria.
* Children with symptoms related to sleep disturbances.
* Children who present episodes of disruptive behaviour.
* Children who may present sensory alterations or cognitive deficits.
* Children whose parents sign the informed consent form.

Exclusion Criteria:

* Present some of the contraindications for treatment with NESA XSIGNAL®: pacemakers, internal haemorrhages, not applying electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and/or phobia of electricity.
* If parents do not sign the informed consent form.
* Presence of uncontrolled convulsions.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality with the Sleep Disturbance Scale for Children (SDSC) | Measurement of change: before treatment (baseline), at two months (end of treatment).
  The Sleep Disturbance Scale for Children (SDSC) will be used. The SDSC is a 26-item scale developed to assess the presence of sleep difficulties in children within the previous six months. The measure is completed by the parent of the child and takes approximately 5-10 min to complete. Item 1 measures the child's average hours of sleep, from 1 ('9 - 11 h') to 5 ('less than 5 h').
Measuring sleep habits with the Children's Sleep Habits Questionnaire scale | Measurement of change: before treatment (baseline), at two months (end of treatment).
  Each scored question is rated on a 3-point scale as occurring "usually" (i.e., 5-7 times within the past week), "sometimes" (i.e., 2-4 times within the past week), or "rarely" (i.e., never or 1 time within the past week).
Change in parent´s sleep quality with the Pittsburgh Sleep Quality Index (PSQI) | Measurement of change: before treatment (baseline), at two months (end of treatment).
  The investigators want to see if there are improvements in the quality, efficiency, and quantity of sleep. The Pittsburgh Sleep Quality Index (PSQI) will be combined to report changes in the patient's sleep quality.
  Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep

SECONDARY OUTCOMES:
Changes to the Register of Disruptive Behaviour Scores with the Aberrant Behavior Checklist (ABC-C) | Measurement of change: before treatment (baseline), at two months (end of treatment).
  The Aberrant Behavior Checklist (ABC-C) is a 58-item rating scale derived by factor analysis, and its five subscales are labelled as follows: I- Irritability (15 items); II- inactivity-isolation (16 items); III- stereotypies (7 items); IV- Hyperactivity, non-compliance (16 items) and V- inappropriate language (4 items). The ABC-C is easy to use, it is completed by an informant such as a teacher, therapist, monitor, parent or other adult who has regular contact with the patient. Each behavioural item is rated on a four-point scale from 0 (not a problem) to 3 (problem is severe).
Change in the stress level of parents with the Change in the stress level of parents | Measurement of change: before treatment (baseline), at two months (end of treatment).
  The Parenting Stress Index-Short Form (PSI-SF) is one of the most commonly used measures of parenting stress both in clinical and research contexts. The PSI-SF is a 36-item, self-report measure with three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (PCDI), and Difficult Child (DC).
  To compute the parental stress score, items 1, 2, 5, 6, 7, 8, 17, and 18 should be reverse scored as follows: (1=5) (2=4) (3=3) (4=2) (5=1). The item scores are then summed. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Change in parental satisfaction with the Parent Satisfaction Questionnaire (PSQ - FS) | Measurement of change: before treatment (baseline), at two months (end of treatment).
  The 19-item PSQ assesses parents' cognitions and perceptions regarding the degree and kind of support they provide to their child following the discovery of sexual abuse. The measure yields a total score and scores on Support and Blame subscales

OTHER OUTCOMES:
Recording of adverse phenomena | From the start of treatment to the end of treatment (2 months)
  The responses experienced by the participant will be observed during the session. As the procedure is sensory imperceptible and easy to handle, it will allow the participant to carry out activities (school/rehabilitation) simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- University of Las Palmas de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parr J. Autism. BMJ Clin Evid. 2010 Jan 7;2010:0322. PMID 21729335
- [Result] Moss AH, Gordon JE, O'Connell A. Impact of sleepwise: an intervention for youth with developmental disabilities and sleep disturbance. J Autism Dev Disord. 2014 Jul;44(7):1695-707. doi: 10.1007/s10803-014-2040-y. PMID 24442795
- [Result] Souders MC, Zavodny S, Eriksen W, Sinko R, Connell J, Kerns C, Schaaf R, Pinto-Martin J. Sleep in Children with Autism Spectrum Disorder. Curr Psychiatry Rep. 2017 Jun;19(6):34. doi: 10.1007/s11920-017-0782-x. PMID 28502070
- [Result] Hirata I, Mohri I, Kato-Nishimura K, Tachibana M, Kuwada A, Kagitani-Shimono K, Ohno Y, Ozono K, Taniike M. Sleep problems are more frequent and associated with problematic behaviors in preschoolers with autism spectrum disorder. Res Dev Disabil. 2016 Feb-Mar;49-50:86-99. doi: 10.1016/j.ridd.2015.11.002. Epub 2015 Dec 10. PMID 26672680